CLINICAL TRIAL: NCT03443440
Title: Delineating Neurocognitive Prognostic Factors Associated With Postoperative Cognitive Dysfunction After General or Neuraxial Anesthesia Utilizing the CogState Brief Battery
Brief Title: Prognostic Factors Associated With Postoperative Cognitive Dysfunction After Surgery
Acronym: POCDCOG
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Kunal Karamchandani, Assistant Professor, Dept. of Anesthesiology & Perioperative Medicine, Milton S. Hershey Medical Center
Other Study IDs: STUDY0000
Record Dates: First submitted 2018-02-13; First posted 2018-02-23 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Neurocognitive Testing — neurocognitive testing, computerized
  Other Names: CogState Brief Battery

SUMMARY:
A longitudinal observational study examining preoperative, intraoperative and postoperative factors associated with Postoperative Cognitive Dysfunction in patients older than the age of 50.

DETAILED DESCRIPTION:
A longitudinal observational study examining factors associated with Postoperative Cognitive Dysfunction (POCD) utilizing a computerized neurocognitive battery. In addition, investigators seek to assess the presence of pre-existing psychiatric disorders and chronic pain to determine their relationship with POCD. The study will seek to compare the rates of POCD in previously published literature with performance on a computerized neurocognitive battery. In addition, the study will seek to determine preoperative, intraoperative and postoperative factors associated with POCD by comparing these variables to performance on a computerized neurocognitive battery.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to perform informed consent
2. Age greater than 50 years old
3. Ability to read and understand English
4. Undergoing elective surgery with general or neuraxial anesthesia

Exclusion Criteria:

1. Patients who do not meet above defined criteria, patients from vulnerable populations (adults unable to consent, pregnant women, prisoners), patients refusing informed consent and participation in the study.
2. A previous history of the following medical conditions: dementia of any kind (vascular dementia, Alzheimer's disease, organic brain disease with documented cognitive deficits, severe traumatic brain injury, Parkinson's disease, senility)
3. Physical impairment impairing their ability to perform neurocognitive testing incl. essential tremor, loss of upper extremity motor function, blindness, or severe hearing loss)

Ages: 50 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult population over the age of 50 years old undergoing general, neuraxial or regional anesthesia for elective surgery.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-06-06 (Actual); Study Completion 2020-06-06 (Actual)

PRIMARY OUTCOMES:
Change in performance on the CogState Brief Battery | Change from baseline on the Cogstate Brief Battery score at postoperative Day 30-40.
  Neurocognitive Test. Detection Task (Score: normal - abnormal), One Card Learning Task (Score: normal - abnormal) One Back Task (Score normal - abnormal) Identification Task (Score normal - Abnormal) Scores are based on normal distributed population data. Scores are measured on a linear scale with no maximum score. Research subjects will also act as their own control based on baseline performance in this longitudinal study.

SECONDARY OUTCOMES:
Change in performance on the Beck Clinical Depression Inventory (BDI) | Change in baseline on the Beck Clinical Depression Inventory at postoperative Day 30-40.
  Test for symptoms of clinical depression. (Scored: 1 to >40 from normal to extreme depression)
Change in performance on the Short-Form McGill Pain Questionnaire (SF-MPQ-2) | Change in baseline on the SF-MPQ-2 at postoperative Day 30-40.
  Test of presence of chronic pain (Scored 0-3(severe)) Validates the sensory component of neuropathic or chronic pain, a visual analog scale (Scored: no pain to worst possible pain) and a Present Pain Intensity (Scored: 0-5 (worst)).
Barthel Index of Activities of Daily Living | Change in baseline on the Barthel Index at postoperative Day 30-40.
  Scale to assess independent function of patient. Components assessing continence, mobility, transfer skills, grooming, hygiene, feeding, bathing, stairs and dressing. (Scored: 0-2, dependent - completely independent) Total Score 0-20 (fully dependent - fully independent)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alosco ML, Spitznagel MB, Strain G, Devlin M, Cohen R, Crosby RD, Mitchell JE, Gunstad J. Pre-operative history of depression and cognitive changes in bariatric surgery patients. Psychol Health Med. 2015;20(7):802-13. doi: 10.1080/13548506.2014.959531. Epub 2014 Sep 15. PMID 25222138
- [Background] Bortolato B, Carvalho AF, McIntyre RS. Cognitive dysfunction in major depressive disorder: a state-of-the-art clinical review. CNS Neurol Disord Drug Targets. 2014;13(10):1804-18. doi: 10.2174/1871527313666141130203823. PMID 25470396
- [Background] Harrington KD, Lim YY, Ames D, Hassenstab J, Rainey-Smith S, Robertson J, Salvado O, Masters CL, Maruff P; AIBL Research Group. Using Robust Normative Data to Investigate the Neuropsychology of Cognitive Aging. Arch Clin Neuropsychol. 2017 Mar 1;32(2):142-154. doi: 10.1093/arclin/acw106. PMID 27932344